CLINICAL TRIAL: NCT07400484
Title: A Study on the Differences in N-CAD Concentration and Brain Function Between Children With Autism Spectrum Disorder and Typically Developing Children
Brief Title: Differences in N-CAD Concentration and Brain Function Between Children With ASD and TD
Status: Recruiting | Type: Observational
Sponsor: Chen Li (Other)
Responsible Party: Sponsor-Investigator, Chen Li, Professor，Director, Children's Hospital of Chongqing Medical University
Organization: Children's Hospital of Chongqing Medical University (Other)
Other Study IDs: DNCBFBCASDTDC
Record Dates: First submitted 2026-01-25; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: ASD
Keywords: ASD; Neural cadherin; Functional Near-infrared Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — 3ml of peripheral blood was collected from the subjects, and the plasma was rapidly separated and frozen in a -80 ℃ refrigerator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ASD: 1. Age at enrollment ≥ 3 years and <5 years;
  2. The diagnosis was made by 2 developmental behavioral pediatricians or child psychiatrists with vice senior titles or above, and the history and clinical manifestations were in line with ASD and ICD-11 diagnostic criteria for ASD.
- TD: Match children with ASD based on age and gender, with normal developmental levels (Gesell DQ ≥ 85).

SUMMARY:
The incidence of autism spectrum disorders is increasing, about 1 / 36. Neural cadherin (NCAD) is closely related to synaptic structure and function. The cdh2 gene encoding NCAD has been shown to be associated with a variety of neurodevelopmental diseases and is one of the six risk genes for ASD. Functional near-infrared spectroscopy (fNIRS) is a neuroimaging technology that uses the principle of near-infrared spectroscopy to detect the functional activation of human cortex. The application of fNIRS to explore the neural mechanism of children with ASD has developed rapidly. It has the advantages of non-invasive, portable, relatively low cost and unlimited physical activity. And for ASD children, their command compliance and self-control are relatively low, so fNIRS is more widely used in ASD children. According to dsm-5 standard, we recruited ASD children and TD children, collected their peripheral blood, and detected the plasma n-cad concentration. At the same time, the resting state of fNIRS of the two groups of children was collected, and the ultra scan monitoring was carried out simultaneously during Gesell assessment. The purpose of this study was to explore the difference of peripheral blood NCAD concentration between preschool ASD children and TD children and the difference of brain function in resting state and social interaction state. And the relationship between the characteristics of brain function and the level of cognitive development in children with ASD.

DETAILED DESCRIPTION:
1. Procedure. Children in ASD group and TD group will complete free physical measurement, blood routine and serum nutrient tests, neuropsychological assessment, and near-infrared brain functional imaging after signing up and giving informed consent. 3ml of peripheral blood was collected from the subjects, and the plasma was rapidly separated and frozen in a -80 ℃ refrigerator. The resting state of ASD and TD children was collected using fNIRS, and the ultra scan monitoring was performed simultaneously during Gesell assessment
2. Demographic questionnaires and clinical data. The demographic questionnaire was completed by the child's primary caregiver, specifying the child's name, sex, and date of birth. Clinical data will be determined from medical records, including relevant dsm-5 diagnosis, disease classification, etc. The
3. Sample size. The sample size was calculated by g*power 3.1. The paired t-test was used to set the effect size d=0.35, α =0.05 (two-sided) Power=0.9， Software calculation showed that 44 cases were needed in each group. Considering the group variability of children and the 10% dropout rate, 49 cases in each group (49 cases in ASD group and 49 cases in TD group) were finally included.
4. Statistical analysis. ① NCAD: the R language 4.5.1 statistical software is used for data analysis. The measurement data conforming to the normal distribution adopts the mean ± standard deviation, and the paired sample t test is used for comparison between groups; The median (quartile) was used for non normally distributed measurement data, and Wilcoxon signed rank test was used for comparison between groups. ② Near infrared: nirspark software was used for data preprocessing, R language 4.5.1 statistical software was used for data analysis, Pearson correlation was used for correlation between channels, and generalized linear model (GLM) or mixed effects model was used for comparison between groups. Multiple linear regression model (adjusting for covariates such as age and gender) was used to explore the association between brain activation and DQ level in children with ASD.
5. ethical issues and data protection. Patients participating in the study will sign an informed consent form. This study was approved by the local ethics committee. . Parents' authorization of patients' health information remained valid until the study was completed. After that, the researcher will delete the private information from the research record.

ELIGIBILITY:
Inclusion Criteria:

1. Age at enrollment ≥ 3 years and <5 years;
2. The diagnosis was made by 2 developmental behavioral pediatricians or child psychiatrists with vice senior titles or above, and the history and clinical manifestations were in line with ASD and ICD-11 diagnostic criteria for ASD; .

Exclusion Criteria:

1. Diagnosis or manifestation of genetic diseases or syndromes related to ASD (such as Rett syndrome);
2. Medical or nervous system diseases affecting growth, development or cognition (such as central nervous system infection, epilepsy, congenital heart disease, etc.);
3. Sensory impairment such as vision or hearing loss;
4. Low birth weight (birth weight <2000 g) or preterm birth (gestational age <37 weeks);
5. Adopted children;
6. Parents refused to sign the informed consent form;
7. Other researchers consider it inappropriate to participate in the study.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: ASD
Sampling Method: Non-Probability Sample
Enrollment: 98 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
N-CAD | Baseline
  NCAD concentration in peripheral blood: N-cadherin (NCAD) in peripheral blood is a calcium dependent cell adhesion molecule, which is mainly involved in cell-cell recognition and adhesion, and is commonly found in nerve tissue, muscle and vascular endothelium. In peripheral blood, the content is very low under normal conditions, but if N-cadherin is detected to be increased, it may be related to tumor metastasis (such as breast cancer, prostate cancer and other epithelial mesenchymal transition), vascular endothelial injury or some neurological diseases. It can be used as a potential biological marker of tumor invasion or vascular abnormalities, but its detection needs to be combined with other indicators to improve the accuracy.
fNIRS | Baseline
  FNIRS (resting state + superscan): functional near infrared spectroscopy (fNIRS) is a noninvasive brain imaging method that detects hemodynamic changes in the cerebral cortex (such as oxygenated hemoglobin and deoxyhemoglobin concentrations) through near-infrared light, thereby indirectly reflecting neural activity. Resting state fNIRS is used to study the spontaneous activity of the brain in the task-free state, and is often used to explore brain functional networks, disease markers (such as mental disorders or neurodegenerative diseases) and individual differences. While fNIRS hyperscanning synchronously records the brain activity of multiple subjects (such as two people interacting), which is used to study the inter brain synchronization in social cognition, cooperation or competition, and reveal the interpersonal neural mechanism. The combination of the two can expand the understanding of brain resting function and social interaction, and is suitable for psychology, neuroscience a

CONTACTS AND LOCATIONS:
Overall Officials: Li Chen, doctor, Study Chair — Children's Hospital of Chongqing Medical University
Locations (1):
- Growth, Development and Mental health of Children and Adolescence Center, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Data is confidential during the study.

REFERENCES:
- [Result] Harrison OJ, Jin X, Hong S, Bahna F, Ahlsen G, Brasch J, Wu Y, Vendome J, Felsovalyi K, Hampton CM, Troyanovsky RB, Ben-Shaul A, Frank J, Troyanovsky SM, Shapiro L, Honig B. The extracellular architecture of adherens junctions revealed by crystal structures of type I cadherins. Structure. 2011 Feb 9;19(2):244-56. doi: 10.1016/j.str.2010.11.016. PMID 21300292
- [Result] Jobsis FF. Noninvasive, infrared monitoring of cerebral and myocardial oxygen sufficiency and circulatory parameters. Science. 1977 Dec 23;198(4323):1264-7. doi: 10.1126/science.929199.
- [Result] Ferrari M, Quaresima V. A brief review on the history of human functional near-infrared spectroscopy (fNIRS) development and fields of application. Neuroimage. 2012 Nov 1;63(2):921-35. doi: 10.1016/j.neuroimage.2012.03.049. Epub 2012 Mar 28. PMID 22510258
- [Result] Liu D, Cao H, Kural KC, Fang Q, Zhang F. Integrative analysis of shared genetic pathogenesis by autism spectrum disorder and obsessive-compulsive disorder. Biosci Rep. 2019 Dec 20;39(12):BSR20191942. doi: 10.1042/BSR20191942. PMID 31808517
- [Result] Christensen DL, Baio J, Van Naarden Braun K, Bilder D, Charles J, Constantino JN, Daniels J, Durkin MS, Fitzgerald RT, Kurzius-Spencer M, Lee LC, Pettygrove S, Robinson C, Schulz E, Wells C, Wingate MS, Zahorodny W, Yeargin-Allsopp M; Centers for Disease Control and Prevention (CDC). Prevalence and Characteristics of Autism Spectrum Disorder Among Children Aged 8 Years--Autism and Developmental Disabilities Monitoring Network, 11 Sites, United States, 2012. MMWR Surveill Summ. 2016 Apr 1;65(3):1-23. doi: 10.15585/mmwr.ss6503a1. PMID 27031587